CLINICAL TRIAL: NCT00266916
Title: Percutaneous Interventions in Adults With Complex Cyanotic Congenital Heart Disease
Brief Title: Percutaneous Interventions in Adults With CHD
Status: Terminated | Type: Observational
Why Stopped: data collection sufficient
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-138
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Last update posted 2007-05-23 (Estimated); Status verified 2007-05

CONDITIONS: Congenital Disorders
Keywords: adult; congenital heart disease; percutaneous occlusion; percutaneous balloon valvotomy; balloon angioplasty; complex cyanotic congenital heart defects (CCHD)
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
The primary objective of this study is to determine the clinical benefits of percutaneous intervention to improve pulmonary blood flow on oxygen saturations, symptoms, exercise tolerance and hematocrit in patients with complex cyanotic congenital heart disease who are not candidates for surgical repair.

DETAILED DESCRIPTION:
This is a single center, retrospective study of adult patients with a diagnosis of un-repaired complex cyanotic congenital heart disease including Eisenmenger's Syndrome, single ventricle, pulmonary atresia with aorticopulmonary collaterals, complete atrio-ventricular canal defects, double inlet left ventricle, heterotaxy syndromes and truncus arteriosus. Patients with surgically placed systemic to pulmonary artery shunts will be included.

Although generally incompatible with adult survival, rare patients with un-operated or palliated complex cyanotic congenital heart defects (CCHD) survive well into adulthood. Symptoms related to poor pulmonary blood flow and/ or increasing pulmonary vascular resistance progress with advancing age. Percutaneous interventions to improve symptoms and relieve hypoxemia have not been previously reported in adult patients with complex cyanotic congenital heart disease. Percutaneous interventions in patients with cyanotic congenital heart disease may be generally broken down into three types: percutaneous occlusion of shunt lesions, percutaneous balloon valvotomy or valvuloplasty, and balloon angioplasty and stenting of vascular structures (1). Percutaneous interventions for occluded or stenotic systemic to pulmonary artery shunts in childhood have been described (2,3). However, procedures to improve pulmonary blood flow in adults with CCHD have not previously been described.

ELIGIBILITY:
Inclusion Criteria:

* greater than 18 years of age
* complex cyanotic heart disease
* oxygen saturation prior to intervention < 90%

Exclusion Criteria:

* those who do not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9
Dates: Start 1996-01; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: Wendy M. Book, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States